CLINICAL TRIAL: NCT03825354
Title: Brief Intervention and Contact (BIC) Program to Manage Suicidal Behaviour: A Pilot Study
Brief Title: Brief Intervention and Contact (BIC) Program
Acronym: BIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Zainab Samaan (Zena), Associate Professor, St. Joseph's Healthcare Hamilton
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Project Number: 5880
Record Dates: First submitted 2019-01-24; First posted 2019-01-31 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2021-09

CONDITIONS: Suicidal Behavior
Keywords: suicide; thoughts; attempts; death; brief intervention; contact
MeSH Terms: conditions — Suicide; Death | interventions — imidazole mustard

STUDY DESIGN:
Intervention Model Description: a randomized study with 1:1 parallel design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief Intervention and contact (BIC) (Experimental): Brief education about suicidal behaviour and follow up contacts for 6 months in addition to treatment as usual. follow up will occur at the following time points post discharge: weeks 1, 2, 4, 6, 8, 12, 16 and 20. this will occur in addition to treatment as usual.
  Interventions: Behavioral: BIC
- control (No Intervention): control will continue treatment as usual which is whatever the clinical team decides upon post discharge. data will be collected on repeated suicidal behaviour through medical records with consent.

INTERVENTIONS:
Behavioral: BIC — World Health Organization, WHO, Brief Intervention and Contact (BIC)
  Arms: Brief Intervention and contact (BIC)

SUMMARY:
Suicide is a significant public health concern and causes approximately 1.5 % of all deaths in the general population in Canada. Suicide is a multi-faceted issue that is often comorbid with psychiatric illness and associated with diverse sociodemographic risk factors. Consequently, there are several domains of suicide risk management. The proposed intervention, the brief intervention, and contact (BIC) model will be tested for feasibility using a pilot pragmatic randomized trial.

DETAILED DESCRIPTION:
Brief contact interventions are distinct from other treatments for suicide and suicidal behaviour, in that the goals include maintaining long-term contact with patients, and through this, provide opportunities for them to re-engage with mental health services when needed. Additionally, brief interventions are not required to be carried out by mental health professionals (i.e. psychiatrists, psychologists, social workers), and they are provided over a structured schedule over a prolonged period post discharge.

The brief intervention and contact (BIC) model followed in this study is based on the BIC model that was utilised by the WHO as part of the Multisite Intervention Study On Suicidal Behaviours (SUPRE-MISS). A sub-project of the SUPRE-MISS study involved the implementation of a brief intervention that included an hour-long information session about suicide and suicidal behaviour around the discharge period, and nine periods of follow up through an in-person visit or phone call to assess the patient's well-being and provide referrals to clinical services as needed. Following implementation, an analysis of the effectiveness of the BIC model in five different countries, Brazil, India, Sri Lanka, Islamic Republic of Iran, and China, outline its potential utility. Compared to patients in the control group, there was a reduction in suicide rates in patients who received the BIC intervention.

This is a pilot study to test the feasibility of implementing the BIC protocol in a large multisite trial. We will, however, provide the objective of the main study to provide an overview of the study and the intended outcomes in addition to the pilot study objectives as below.

Study question and hypothesis of the main study:

For patients with suicidal behaviour admitted to inpatient units of acute and tertiary hospitals, does the addition of a brief intervention and contact program decrease suicide re-attempts, reduce depressive symptoms, improve social connectivity, and reduce further ER visits, compared to treatment as usual after 18 months of follow-up? The pilot study will be for 6 months only. We hypothesize that brief intervention and contact is an effective intervention for reducing suicidal behaviour in patients who have attempted suicide.

The intervention:

Patients in the intervention group will receive the BIC intervention, alongside treatment as usual. BIC consists of a 1-hour information session about the epidemiology and presentation of suicide and suicidal behaviour at the time of discharge, along with follow-up with patients at 1, 2, 4, 6 weeks, and 3, 4, 5, and 6 months. The intention of the frequency of follow up is to increase the time between follow up visits as per the original protocol and eventually discontinue. Follow-up contact will involve assessing how patients feel and whether they need additional support. The WHO protocol that contains all questionnaires to be used for follow-up is attached to this protocol.

The control:

Patients in the control group will receive treatment as usual. Pilot Study Objectives

Primary objectives:

The main goal of pilot phase is to enhance the success of the full trial by testing the feasibility of conducting a randomized controlled trial to assess the effectiveness of a brief intervention and contact program for suicide delivered through a face to face, phone or text-based intervention in addition to treatment as usual to reduce suicide attempts, depressive symptoms and ER visits, and improve social connectivity.

The pilot primary objectives are therefore summarized after Thabane and colleagues (cite the ref here):

1. Assess the feasibility of the study process in terms of recruitment, retention, number of follow-ups completed, and data completion
2. Assess resources needed including the use of mobile phones for contacting patients, interview spaces for initial intake questionnaire and consent processes.

Pilot study secondary objectives

1. Assess reduction in subsequent suicide attempts and completed suicides through access to medical records over 6 months post discharge
2. Assess the change in depressive symptoms using the Beck Depression Inventory between and within the intervention and control groups
3. Explore the change in sense of social connectivity and social support using the Bille-Brahe Social Support Questionnaire, the Sarason Social Support Questionnaire (short form), and two questions pertaining to the places and activities the patient engages in most often between and within the intervention and control groups
4. Assess the reduction in ER visits between and within the intervention and control groups

ELIGIBILITY:
Inclusion Criteria:

* All patients with a previous suicide attempt or expressed any suicidal behaviour who are admitted to inpatient psychiatric wards will be asked to participate in this study, with no upper age limit, sex or gender restriction.
* No restrictions will be placed on the patients' diagnoses or comorbidities, although all diagnoses will be documented.
* Patients in inpatient units and receiving treatment for comorbid psychiatric illnesses and/or their suicidal behaviour as per usual care including medication, individual or group psychotherapies and other treatment modalities are eligible to participate in the study.
* All participants must be able to provide written informed consent and can be reached through phone calls and/or text messages or in-person visits to the hospital site.

Exclusion Criteria:

* We will exclude patients who are unable to understand written and spoken English, as the research staff/clinicians delivering the intervention are limited to English-speaking populations.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | 6 months
  The percentage of potential participants agree to consent to the study
Retention rate | 6 months
  The percentage of participants who completes the study
Data completion rate | 6 months
  the percentage of participants who complete all study questionnaires and follow up contacts

SECONDARY OUTCOMES:
The number of suicidal behaviour events | 6 months
  The number of documented suicidal behaviour events including ideas, attempts and completion

CONTACTS AND LOCATIONS:
Overall Officials: z Samaan, MD/PhD, Principal Investigator — McMaster University
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Soni D, Panesar B, Dufort A, Guan L, Lee J, Waldern D, Hathaway S, Sanger N, Stacey S, Minuzzi L, Thabane L, Samaan Z. Recruitment rates, retention rates, and follow-up completion in a Brief Intervention and Contact trial for suicidal behavior: a feasibility study. Pilot Feasibility Stud. 2025 Apr 16;11(1):50. doi: 10.1186/s40814-025-01635-3. PMID 40241209